CLINICAL TRIAL: NCT05463237
Title: The Relation Between Visceral Adipokines Gestational Diabetes Mellitus
Brief Title: Comparison of Visceral Adipokines Visfatin, Vaspin and Omentin Levels in Gestational Diabetes Mellitus Pregnant Women
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, associate professor, Siirt University
Other Study IDs: SiirtUNI
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Gestational Diabetes; Obesity; Visceral Obesity
MeSH Terms: conditions — Diabetes, Gestational; Obesity; Obesity, Abdominal | interventions — Glucose Tolerance Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with gestational diabetes(n:87): Visceral adipokine level will be examined in pregnant women with gestational diabetes.
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: Blood sample
- Control group pregnant (n:87): Visceral adipokine level will be examined in pregnant women with normal pregnant .
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test — oral glucose tolerance test (OGTT) used for the diagnosis of gestational diabetes mellitus between 24-28 weeks of gestation
Diagnostic Test: Blood sample — Measurement of blood Visfatin, Vaspin and Omentin levels in pregnant women with diabetes

SUMMARY:
The prevalence of maternal obesity is increasing rapidly worldwide and constitutes an important obstetric problem that increases mortality and morbidity in both mothers and infants. Obese women are prone to pregnancy complications such as gestational diabetes mellitus (GDM), and children of obese mothers are more likely to develop cardiovascular and metabolic disease later in life. The risk of developing GDM in obese pregnants is 1.3-3.8 times higher than in pregnant women with a normal body mass index, and approximately 70% of women with GDM remain at risk of developing type 2 diabetes until 28 years postpartum. Gestational diabetes mellitus (GDM) affects approximately 6% of pregnant women and its prevalence is increasing in parallel with the obesity epidemic. GDM is associated with an increased risk of adverse pregnancy outcomes, including macrosomia, preterm delivery, neonatal hypoglycemia, neonatal jaundice, and congenital anomalies. It is also associated with a higher incidence of type 2 diabetes mellitus after birth. It is known that visceral adipose tissue increases in obese women. It is thought that there is a relationship between visceral adipose tissue increase and diabetes. In this study, the levels of new adipocytokines such as Visfatin, Vaspin and Omentin secreted from visceral adipose tissue in patients diagnosed with GDM will be measured.

DETAILED DESCRIPTION:
The investigators aim in this study the levels of Visfatin, Vaspin and Omentin secreted from this tissue in pregnant women diagnosed with GDM by oral glucose tolerance test (OGTT) between 24-28 weeks of gestation and to determine if there is a relationship between these parameters. For this purpose, , and 87 pregnant women with gestational diabetes diagnosed at 24-28 weeks from the same patient group will be included in the study. . The same number of non-GDM control group pregnant women will also be included in the study at 24-28 weeks. Age, gestational week, pregnancy history (gravida, parity, abortion, missed, ectopic), medical history, preconceptional BMI, current BMI, triglyceride, VLDL, HDL, LDL, cholesterol, HOMA-IR, C-peptide, insulin, Hba1c levels will be saved. In the 2nd trimester, between 24-26 weeks, OGTT will be performed on the patients and the results will be recorded. Visfatin, Vaspin and Omentin levels will be checked and recorded in patients diagnosed with GDM.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* At the 2.st trimester of pregnancy

Exclusion Criteria:

* History of with diabetes mellitus
* Morbidly obese pregnants
* History of abdomen liposuction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women over the age of 18 who are in the first trimester of pregnancy and are not diagnosed with diabetes
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
24-28. Visceral Adipokine Levels in Pregnant Women with Gestational Diabetes Between Weeks | Between 24-28 weeks of pregnancy, (an average of 6 months)
  VASPIN, VISFATIN, OMENTIN levels will be measured in patients with gestational diabetic,

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Assoc.Prof, Study Director — Siirt University Medical Faculty Obstetrics and Gynecology Departmant; Şerif Aksin, Study Director — Siirt Üniversity Medical Faculty Obstetrics and Gynecology Department
Locations (1):
- Siirt Üniversity Medical Faculty, Siirt, Turkey (Türkiye)